CLINICAL TRIAL: NCT04643340
Title: Functional Imaging During Subliminal Perception
Brief Title: Imaging During Subliminal Perception
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-00483
Record Dates: First submitted 2020-11-16; First posted 2020-11-25 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: functional MRI; subliminal perception; EEG; neurofeedback; attention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- active group 1: This group will train the insular cortex by real-time fMRI
  Interventions: Other: real-time fMRI
- active group 2: This group will train the visual cortex by real-time fMRI
  Interventions: Other: real-time fMRI
- sham: This group will only train the insula by a particular strategy

INTERVENTIONS:
Other: real-time fMRI — Brain regions can be trained, i.e. fMRI activity can be actively modulated online by humans, using rt-fMRI (Bruhl, Scherpiet et al. 2014, Bruhl 2015, Emmert, Kopel et al. 2016).
  Groups: active group 1; active group 2

SUMMARY:
Subliminal perception of visual stimuli can be studied with functional brain imaging, e.g. with functional magnetic resonance imaging (fMRI). However, it is unclear how subliminal perception affects connectivity in the brain.

Further, it is not known if real-time (rt) fMRI neurofeedback of brain areas involved in subliminal perception can lead to supra-threshold perception.

For attention tasks, the investigators hypothesize that functional connectivity strength is mediated by the insular cortex during both supra-threshold and subliminal perception.

Additionally, the investigators hypothesize that rt-fMRI neurofeedback training should alter neuronal and behavioral responses.

DETAILED DESCRIPTION:
In this project, using healthy adults, the investigators have 2 aims:

1. Apply electroencephalography (EEG) and fMRI before and after rt-fMRI neurofeedback during attention tasks to identify brain regions involved in subliminal and supraliminal perception.
2. Apply functional connectivity analyses during these tasks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (> 18 < 80 years), which can read and sign the informed consent form
* Male and female
* Right-handed

Exclusion Criteria:

* metallic items in the body (i.e. eye splinter, MR incompatible implants)
* pacemaker
* claustrophobia
* pregnant participants
* participants suffering from a degenerative disorder of the Central Nervous System, such as Stroke, Multiple Sclerosis, Parkinson's Disease, Alzheimer's Disease and Huntington's Disease and with major psychiatric disorders such as schizophrenia, depression, or anxiety disorder
* Drug intake (psychopharmaca)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
fMRI during supra-threshold and subliminal perception | 2020 - 2022
rt-fMRI activity | 2020 - 2022
  rt-fMRI activity: fMRI signal changes during repetitive real time fMRI based training

SECONDARY OUTCOMES:
Functional connectivity | 2020 - 2022
  Examination of fMRI signal dependencies (coherence) between brain regions.
EEG activity | 2020 - 2022
  EEG activity: Event related potentials and spectral band power for different trial types
fMRI task performance | 2020 - 2022
  Reaction time and accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Lars Michels, PhD, Principal Investigator — University Hospital, Zürich
Locations (1):
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Raw imaging data can be shared with other groups (outside of the USZ), e.g. for replication purpose.

REFERENCES:
- See also: SNF database — http://p3.snf.ch/project-182803